CLINICAL TRIAL: NCT05335005
Title: A Study to Evaluate Safety and Tolerability of Co-administration of MK-2060 and Clopidogrel in Participants With End-Stage Renal Disease on Hemodialysis
Brief Title: MK-2060 and Clopidogrel Co-administration Safety and Tolerability Study in Participants With End-Stage Renal Disease (ESRD) (MK-2060-008)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2060-008; MK-2060-008 (Other: Merck); 2021-005333-17 (EudraCT Number)
Record Dates: First submitted 2022-04-12; First posted 2022-04-19 (Actual); Results first posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-07

CONDITIONS: End-Stage Renal Disease; Kidney Failure, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MK-2060 (Experimental): Participants continued their established background therapy of daily 75 mg clopidogrel for 2 weeks (days -14 to 0). Participants then continued background therapy while receiving 25 mg MK-2060 intravenous (IV) infusion on days 1, 3, 5, and 8.
  Interventions: Drug: MK-2060

INTERVENTIONS:
Drug: MK-2060 — MK-2060 administered via IV infusion

SUMMARY:
MK-2060 is being developed for prevention of thrombotic complications in end-stage renal disease (ESRD). The purpose of this study is to conduct a preliminary evaluation of the safety and tolerability of MK-2060 treatment in combination with a commonly used P2Y12 receptor inhibitor, clopidogrel, in ESRD patients.

ELIGIBILITY:
Inclusion Criteria:

* Has End-Stage Renal Disease (ESRD) maintained on stable outpatient hemodialysis (HD) regimen at a healthcare center for > 3 months prior to dosing.
* On HD regimen at least 3 times per week for a minimum of 3 hours per dialysis session, using a complication-free well-maintained AV fistula or AV graft.
* Is taking clopidogrel for a minimum of 2 weeks prior to the first dosing of MK-2060 administration.
* Has a Body Mass Index (BMI) ≥ 18 and ≤ 45 kg/m^2.

Exclusion Criteria:

* History of cancer (malignancy), including adenocarcinoma, except adequately treated nonmelanomatous skin carcinoma or carcinoma in situ of the cervix or other malignancies that have been successfully treated with appropriate follow up.
* Has a history of deep vein thrombosis or pulmonary embolism.
* Has a history of gastrointestinal (GI) bleeding, duodenal polyps or gastric ulcer in the last 5 years or severe hemorrhoidal bleed in last 3 months prior to screening.
* Is positive for hepatitis B surface antigen or human immunodeficiency virus (HIV).
* Has ongoing anticoagulant therapy or antiplatelet therapy, not including clopidogrel. Intradialytic heparin is permitted.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2023-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharpe & Dohme LLC
Locations (3):
- Genesis Clinical Research, LLC ( Site 0003), Tampa, Florida, United States
- Hadassah Medical Center-Clinical Reaserch Unit ( Site 0002), Jerusalem, Israel
- ARENSIA Exploratory Medicine-Clinical Nephrology Hospital "Carol Davila" ( Site 0001), Bucharest, București, Romania

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MK-2060
Started | 12
Completed | 11
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | MK-2060
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.3 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experience One or More Bleeding Related Adverse Events (AE)
Description: Bleeding related AEs include any sign or symptom of bleeding, even if not requiring intervention by a medical/healthcare professional, as well as clinically-relevant non major bleeding or major bleeding.
Time Frame: Up to approximately 104 days
Population: The analysis population included all participants who received ≥1 dose of MK-2060.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-2060
Number analyzed (Participants) | 12
Participants | 0

2. Primary Outcome: Number of Participants Who Experience One or More AEs
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Time Frame: Up to approximately 104 days
Population: The analysis population included all participants who received ≥1 dose of MK-2060.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-2060
Number analyzed (Participants) | 12
Participants | 6

3. Primary Outcome: Number of Participants Who Discontinue Study Intervention Due to an AE
Description: as for outcome 2
Time Frame: Up to approximately 8 days
Population: The analysis population included all participants who received ≥1 dose of MK-2060.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-2060
Number analyzed (Participants) | 12
Participants | 0

4. Secondary Outcome: Area Under the Concentration-Time Curve From 0 to 168 Hours (AUC0-168) of MK-2060
Description: The AUC0-168 was defined as the area under the concentration-time curve of MK-2060 in plasma from time zero to 168 hours after administration. The Week 1 value is the extrapolated value using data up to 48 hours postdose Day 1, with the "Partial area" option in WinNonlin software using a Start time of 0 hours and an End time of 168 hours. Week 2 value included data for Day 8: predose, and 1, 12, 24, 48, 96, and 168 hours postdose.
Time Frame: Day 1: predose, and 1, 12, 24, and 48 hours postdose. Day 8: predose, and 1, 12, 24, 48, 96, and 168 hours postdose.
Population: The analysis population included all participants who received ≥1 dose of MK-2060 and who complied with the protocol sufficiently to ensure that the data are likely to exhibit the effects of treatment according to the underlying scientific model.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nmol/L
Arm/Group | MK-2060
Number analyzed (Participants) | 12
hour*nmol/L
  Week 1 | 2040 (27.5)
  Week 2 | 9060 (40.5)

5. Secondary Outcome: Maximum Plasma Concentration (Cmax) of MK-2060
Description: Cmax was defined as the maximum concentration of MK-2060 observed in plasma after administration. Week 2 value included data for Day 8: predose and 1, 12, 24, 48, 96, and 168 hours postdose.
Time Frame: Day 1: predose, and 1, 12, and 48 hours postdose. Day 8: predose, and 1, 12, and 24 hours postdose; and once daily on Days 10, 12, 15, 21, 29, 35, 49, 67, and 104.
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | MK-2060
Number analyzed (Participants) | 12
nmol/L
  Week 1 | 29.7 (19.9)
  Week 2 | 87.6 (24.2)

6. Secondary Outcome: Plasma Concentration at 168 Hours (C168) of MK-2060
Description: C168 was defined as the concentration of MK-2060 observed in plasma 168 hours after administration. Week 2 value included data for Day 8: 168 hours postdose.
Time Frame: Days 1 and 8: 168 hours post-dose
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | MK-2060
Number analyzed (Participants) | 12
nmol/L
  Week 1 | 43.1 (26.7)
  Week 2 | 34.3 (66.2)

7. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of MK-2060
Description: Tmax was defined as the time required to reach the maximum concentration of MK-2060 observed in plasma after administration. Week 2 value included data for Day 8: predose and 1, 12, 24, 48, 96, and 168 hours postdose.
Time Frame: as for outcome 5
Population: as for outcome 4
Measure: Median (Full Range); unit: Hours
Arm/Group | MK-2060
Number analyzed (Participants) | 12
Hours
  Week 1 | 1.03 [0.75 to 1.25]
  Week 2 | 1.07 [0.90 to 12.00]

8. Secondary Outcome: Terminal Half Life (t1/2) of MK-2060
Description: T1/2 was defined as the time required to divide the MK-2060 plasma concentration by two after reaching pseudo-equilibrium.
Time Frame: Day 8: predose, and 1, 12, and 24 hours postdose. Once daily on Days 10, 12, 15, 21, 29, 35, 49, 67, and 104.
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | MK-2060
Number analyzed (Participants) | 11
Hours | 402 (31.5)

9. Secondary Outcome: Clearance at Steady State (CLss) of MK-2060
Description: CLss was defined as the volume of plasma from which MK-2060 was eliminated per unit time following administration, once at steady state.
Time Frame: Day 8: predose, and 1, 12, and 24 hours postdose. Once daily on Days 10, 12, 15, 21, 29, 35, 49, 67, and 104.
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hour
Arm/Group | MK-2060
Number analyzed (Participants) | 11
L/hour | 0.0170 (25.6)

10. Secondary Outcome: Apparent Volume of Distribution at Steady State (Vss) of MK-2060
Description: Vss was defined as the volume of plasma that would be necessary to contain the total amount of administered MK-2060 at the same concentration that MK-2060 was observed in the blood plasma after reaching steady state.
Time Frame: Day 8: predose, and 1, 12, and 24 hours postdose. Once daily on Days 10, 12, 15, 21, 29, 35, 49, 67, and 104.
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | MK-2060
Number analyzed (Participants) | 11
Liters | 6.34 (33.3)

11. Secondary Outcome: Time to Hemostasis Following MK-2060 Treatment
Description: Time to hemostasis is assessed by measuring the time that pressure is held from removal of dialysis catheters from the dialysis access site [i.e., arteriovenous (AV) fistula or AV graft] until adequate hemostasis has been obtained for both the arterial and venous sites.
Time Frame: Up to approximately 15 days
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: Minutes
Arm/Group | MK-2060
Number analyzed (Participants) | 12
Minutes | 11.0 [6.97 to 15.1]

ADVERSE EVENTS:
Time Frame: Run-in (Clopidogrel 75 mg) arm: Approximately 14 days MK-2060 25 mg IV/Clopidogrel 75 mg arm: Up to approximately 108 days
Groups:
- Run-in (Clopidogrel 75 mg): Participants continued their established background therapy of daily 75 mg clopidogrel for 2 weeks (days -14 to 0).
- MK-2060 25 mg IV/Clopidogrel 75 mg: In addition to standard background therapy of 75 mg clopidogrel, participants received 25 mg MK-2060 intravenous (IV) infusion on days 1, 3, 5, and 8.
Arm/Group | Run-in (Clopidogrel 75 mg) | MK-2060 25 mg IV/Clopidogrel 75 mg
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 3/12
Other Adverse Events (participants affected / at risk) | 1/12 | 5/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Run-in (Clopidogrel 75 mg) (N=12) | MK-2060 25 mg IV/Clopidogrel 75 mg (N=12)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Run-in (Clopidogrel 75 mg) (N=12) | MK-2060 25 mg IV/Clopidogrel 75 mg (N=12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Renal hypertension (Renal and urinary disorders) | 0 (0) | 1 (2)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-09): https://cdn.clinicaltrials.gov/large-docs/05/NCT05335005/Prot_SAP_000.pdf